CLINICAL TRIAL: NCT02738190
Title: Albumin vs. Plasma for PEdiAtric pRiming Trial
Acronym: APPEAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, MD, FESC, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APPEAR
Record Dates: First submitted 2016-03-15; First posted 2016-04-14 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Hemorrhage
Keywords: albumin; fresh frozen plasma; extracorporeal circulation; cardiovascular surgery; pediatric population
MeSH Terms: conditions — Hemorrhage | interventions — Albumins; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albumin (Active Comparator): 5% Albumin to be added to the priming solution composed of concentrated red cells to reach a target of 28-30% hematocrit and albumin to reach the standard volume administered to these patients (400 ml)
  Interventions: Drug: Albumin
- Fresh Frozen Plasma (Active Comparator): Fresh Frozen Plasma to be added to the priming solution composed of concentrated red cells to reach a target of 28-30% hematocrit and plasma to reach the standard volume administered to these patients (400 ml)
  Interventions: Biological: Fresh Frozen Plasma

INTERVENTIONS:
Drug: Albumin — Albumin 5% added to blood priming solution
  Other Names: Albumina; Human Albumin
  Arms: Albumin
Biological: Fresh Frozen Plasma — Fresh Frozen Plasma added to blood priming solution
  Arms: Fresh Frozen Plasma

SUMMARY:
This is a randomized controlled trial that compares two different priming composition (albumin vs. fresh frozen plasma) for extracorporeal circulation of pediatric patients under 10 kg of weight. The two approaches are both employed at the moment but there is actually no evidence on the superiority of one over the other. This study is aimed to test the hypothesis that Albumin is superior to fresh frozen plasma in terms of minor bleeding and transfusional requirements.

DETAILED DESCRIPTION:
Extracorporeal circulation (ECC) in neonates and infants undergoing cardiac surgery for the correction or palliation of cardiac defects is characterized by temperature variation, activation of coagulation and inflammatory cascades, hemodilution.

An excessive dilution of circulating mass determines a variation in colloid-oncotic pressure (COP) that, together with hydrostatic pressure, induces liquids exchange between interstitial space and plasma. COP variation together with inflammatory response due to extracorporeal circulation and temperature variation is the main determinant of interstitial and pulmonary edema occurrence. Intravascular albumin is responsible for 80% for the COP. Golab et al. randomized a population of neonates and infants undergoing to pediatric cardiac surgery procedures in order to reach two different targets of COP through administration of different albumin amounts. His results didn't show significant differences for primary and secondary endpoints except for postoperative ventilation duration.

Trials on adult patients undergoing cardiac surgery haven't showed differences in bleeding when varying colloid solution employed. Albumin is preferred to artificial colloids due to reduced risk of anaphylactic reactions and for its capacity to maintain COP.

Hemodilution is associated to a reduction in hematocrit, platelet count, fibrinogen and other coagulation factor concentration. Solutions employed for ECC (Extracorporeal Circulation) circuits priming also contain components that could impair hemostasis.

In order to reduce the negative effects on the coagulation, many centers for pediatric surgery employ fresh frozen plasma (FFP) for priming solution. Oliver et al randomized a population of 51 cardiopathic, acyanotic children under 10 kg of weight to receive either albumin or FFP as ECC priming. The authors showed a reduction of postoperative bleeding in the group receiving FFP. No significant differences were detected in postoperative coagulation tests. Other studies with small cohorts weren't able to detect significant differences between the two regimens applied by Oliver and colleagues.

Currently the patients receiving blood priming are treated with either FFP or albumin in order to maintain a correct COP. Comparative studies are very limited by small populations and haven't yet provided definitive conclusions about eventual superiority of one regimen over another.

This is a randomized controlled trial that compares the employment of 5% Albumin (ALB group) versus Fresh Frozen Plasma (FFP group) for priming as per standard protocol of extracorporeal circulation procedure. No modifications to the normal clinical management of the patient are planned. The primary endpoint is to reduce postoperative bleeding (registered as ml/kg in the first 12 postoperative hours). The secondary endpoints are to reduce transfusional requirements for all the blood products (packed red cells, fresh frozen plasma and platelets registered as ml/kg from the beginning of the extracorporeal circulation for up to 48 hours from the termination of the surgery), ventilation support and hospital stay duration. Safety endpoint is represented by the percentage of thromboembolic complications (stroke, peripheric, pulmonary and mesenteric thromboembolisms). Both the treatments employed in this trial are to be considered standard.

ELIGIBILITY:
Inclusion Criteria:

* weight under 10 kg
* cardiovascular surgery procedure with extracorporeal circulation
* need for hematic priming solution
* elective surgery
* informed consent signed

Exclusion Criteria:

* congenital disorders of coagulation system
* emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Volume of postoperative bleeding | 24 hours
  Postoperative bleeding in ml/kg, as measured by chest drainage

SECONDARY OUTCOMES:
Number of units of blood components transfused | 48 hours
  All kind of blood products (packed red cells, fresh frozen plasma, platelet concentrate) transfused from the extracorporeal circulation beginning
Hours on artificial ventilation | hours until extubation, an average of 72 hours
  Artificial ventilation duration from the ICU admission till extubation
Days of hospital stay | days until discharge, an average of 10 days
  Hospital stay duration from ICU admission till discharge
Thromboembolic complications | Postoperative hospital stay until discharge, an average of 10 days
  All kind of thromboembolic complication (peripheric, pulmonary, mesenteric) from ICU admission till discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, FESC, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weil MH, Henning RJ, Puri VK. Colloid oncotic pressure: clinical significance. Crit Care Med. 1979 Mar;7(3):113-6. doi: 10.1097/00003246-197903000-00006. No abstract available. PMID 436426
- [Background] Golab HD, Scohy TV, de Jong PL, Kissler J, Takkenberg JJ, Bogers AJ. Relevance of colloid oncotic pressure regulation during neonatal and infant cardiopulmonary bypass: a prospective randomized study. Eur J Cardiothorac Surg. 2011 Jun;39(6):886-91. doi: 10.1016/j.ejcts.2010.09.040. Epub 2010 Nov 5. PMID 21055963
- [Background] Chandler WL. Effects of hemodilution, blood loss, and consumption on hemostatic factor levels during cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2005 Aug;19(4):459-67. doi: 10.1053/j.jvca.2004.11.046. PMID 16085250
- [Background] Oliver WC Jr, Beynen FM, Nuttall GA, Schroeder DR, Ereth MH, Dearani JA, Puga FJ. Blood loss in infants and children for open heart operations: albumin 5% versus fresh-frozen plasma in the prime. Ann Thorac Surg. 2003 May;75(5):1506-12. doi: 10.1016/s0003-4975(02)04991-3. PMID 12735570
- [Background] McCall MM, Blackwell MM, Smyre JT, Sistino JJ, Acsell JR, Dorman BH, Bradley SM. Fresh frozen plasma in the pediatric pump prime: a prospective, randomized trial. Ann Thorac Surg. 2004 Mar;77(3):983-7; discussion 987. doi: 10.1016/j.athoracsur.2003.09.030. PMID 14992912
- [Derived] Bianchi P, Cotza M, Beccaris C, Silvetti S, Isgro G, Pome G, Giamberti A, Ranucci M; Surgical and Clinical Outcome REsearch (SCORE) group. Early or late fresh frozen plasma administration in newborns and small infants undergoing cardiac surgery: the APPEAR randomized trial. Br J Anaesth. 2017 May 1;118(5):788-796. doi: 10.1093/bja/aex069. PMID 28510741